CLINICAL TRIAL: NCT07368075
Title: Comparison Of Post Operative Analgesic Effectiveness Of Ropivacane Plus Dexamethasone And Ropivacane Plus Dexmedetomidine In Trans Abdominal Plane Block In Stoma Reversal Under General Anesthesia
Brief Title: To Compare Post-op Analgesic Effectiveness of Ropivicaine+Dexamethasone and Ropivacane+Dexmetomidine in TAP Block in Stoma Reversal Under GA in Terms of Duration of Analgesia.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sahiwal medical college sahiwal (Other Government)
Responsible Party: Principal Investigator, Mudassar Ali, Resident Anaesthetist, Sahiwal medical college sahiwal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 213/IRB
Record Dates: First submitted 2026-01-15; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Analgesia; Opioid Sparing Anaesthesia; Hypotension, Controlled; Bradycardia; Stoma Reversal Procedure
MeSH Terms: conditions — Hypotension; Bradycardia

STUDY DESIGN:
Intervention Model Description: Group I patients will receive TAP block with 20 mL 0.25% Rupivacane plus dexamethasone 4 mg at the end of surgery on surgical side. Group II patients will receive 20 mL of 0.25% ropivacaine plus dexmedetomidine 0.25ug/kg body weight at the end of surgery on surgical side
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Ropivacaine+Dexamethasone (Other): patients will receive TAP block with 20 mL 0.25% Rupivacane+dexamethasone 4 mg
  Interventions: Drug: TAP Block with Ropivacaine+Dexamethasone
- Group Ropivacaine+Dexmedetomidine (Other): patients will receive TAP Block with 20 mL of 0.25% ropivicaine+dexmedetomidine 0.25ug/kg
  Interventions: Drug: TAP Block with Ropivacaine+Dexmedetomidine

INTERVENTIONS:
Drug: TAP Block with Ropivacaine+Dexamethasone — With the patient with proper positioning the skin will be disinfected and the transducer positioned. A needle is placed deep to the fascia separating the internal oblique muscle from the transversus abdominis muscle. The needle entry point will be anesthetized with 20 mL 0.25% Rupivacane plus dexamethasone 4 mg. The local anesthetic spreads in this plane, blocking the sensory nerves (like iliohypogastric and ilioinguinal) that run along the abdominal wall.
  Arms: Group Ropivacaine+Dexamethasone
Drug: TAP Block with Ropivacaine+Dexmedetomidine — With the patient with proper positioning the skin will be disinfected and the transducer positioned. A needle is placed deep to the fascia separating the internal oblique muscle from the transversus abdominis muscle. The needle entry point will be anesthetized with 20 mL 0.25% Rupivacane plus dexamedetomidine 0.25ug/kg. The local anesthetic spreads in this plane, blocking the sensory nerves (like iliohypogastric and ilioinguinal) that run along the abdominal wall
  Arms: Group Ropivacaine+Dexmedetomidine

SUMMARY:
Controlling pain is of major concern in intra-operative as well as post-operative period inpatients undergoing all surgeries especially abdominal surgeries.Adequate pain control in post-operative period directly effect patient's recovery and shortens the patient hospital stay consequently decreasing burden on health facilities. Inadequate pain control may affect quality of life and increases patient's morbidity and mortality and is a considerable problem worldwide.

Different modalities for pain control are used in post-operative period. Opioids are main stay of treatment in post-operative period but has significant side effect profile like dependence, nausea & vomiting. Regional blocks like TAP (Trans Abdominal Plane) are now a days being used as post operative analgesia in abdominal surgeries.

The randomized control trial of Comparison of Ropivacane 0.25% plus Dexamethasone and Ropivacane 0.25% plus Dexmedetomedine will be conducted at department of anaesthesia of Sahiwal teaching hospital Sahiwal for 12 months. 86 patients meeting the inclusion criteria will be categorized into two different groups using computer-generated random number table. All patients will undergo a pre-operative assessment on the day before surgery. Both Group will receive TAP block with studied drugs at the end of surgery. After surgery patient will be shifted to post-surgical ward and will be assessed for pain using visual analogue scale (VAS) and data will be collected and analyzed using Statistical Package for the Social Sciences (SPSS) version 26. Quantitative variable will be presented with mean± SD. Comparison of quantitative variable between groups will be done using independent sample-t-test. Comparison of qualitative variable like (opioid sparing effect Nausea,vomiting,Bradycardia,Hypotension) will be presented with frequency and percentages. Data will be stratified on the basis of gender and age. Post-stratification chi-square test will be used to compare both groups for opioid sparing effect in each stratum with p-value≤0.05 as significant

DETAILED DESCRIPTION:
After approval from hospital ethical committee and obtaining informed written consent from every patient, patient fulfilling the criteria of inclusion, demographic statics. Patients will be randomly allocated into two groups using a computer-generated random number table. All patients will undergo a per-operative assessment a day before surgery. They will be per-medicated with oral midazolam 0.05 mg/kg 2 h before surgery. Ultrasound machine SonoScape model S11-plus with linear probe with code L741 and frequency range of 5-10 MHz will be used for ultrasound guidance and 25G Quinkes' lumbar puncture needle will be used for administration of dose. Group I patients will receive TAP block with 20 mL 0.25% Rupivacane plus dexamethasone 4 mg at the end of surgery on surgical side. Group II patients will receive 20 mL of 0.25% ropivicaine plus dexmedetomidine 0.25ug/kg body weight at the end of surgery on surgical side. The person who will prepare the study drugs will not participate in the data collection. Anaesthesia will be induced with propofol 2-2.5 mg/kg intravenous (IV) and 0.1mg/kg intravenous (IV). Tracheal intubation will be facilitated by succinylcholine 1.5 mg/kg IV. Anaesthesia will be maintained with isoflurane 0.6 MAC, 60% nitrous oxide, 40% oxygen, atracurium 0.5mg/kg bolus followed by 0.15mg/kg maintenance dose every 30 mints until completion of surgery. Patients Intraoperative monitoring will include electrocardiogram,non-invasive blood pressure at 5 min intervals, oxygen saturation, end-tidal carbon dioxide and nasopharyngeal temperature. Patients will be ventilated by intermittent positive pressure ventilation using a circle system to maintain normocapnia. Heart rate (HR) and mean arterial pressure (MAP) will be maintained within 20% of the pre-operative value. Hypotension (MAP <20% of the baseline or <65 mmHg) will be treated with infusion of normal saline and if required injection phenylephrine boluses IV. Bradycardia (HR <50 beats/min) will be treated with IV atropine 10 µg/kg bolus in both intraoperative and post-operative period. All patients will receive paracetamol 10 mg/kg IV and ondansetron 0.1 mg/kg IV ½ hour before the completion of surgery. At the end of surgery, residual neuromuscular block will be antagonized with 0.04mg/kg of neostigmine and 0.01 mg/kg glycopyrrolate IV. Tracheal extubation will be performed on meeting the standard criteria for extubation. Patients will be shifted to post anaesthesia care unit (PACU) where resident anaesthesia doctor and trained nursing staff 11 unaware of the studied drug given to the patient will assess patients for pain using visual analogue scale (VAS, 0 score correspond to no pain and 10 score to the worst pain).The time will be noted to first request of analgesia (the time interval between the TAP block done at skin closure and the first request to analgesia at vas 4 or more).Postoperative hemodynamic will be assessed every 30mints for first 4 h then 2 hourly for next 24 hr. Inj nalbuphine 0.1mg/kg intravenously will be given on patient required basis as Rescue drug. Total opioid consumption per 24 hours in both groups in term of mg will be noted.

The incidence of postoperative complication of studied drugs will be noted i.e., Bradycardia,hypotension , Nausea and Vomiting for 24 h postoperatively. The data will be collected through structured questionnaire attached as annexure.

ELIGIBILITY:
Inclusion Criteria:

1. Age limit: 18-60 years
2. Gender of patient i.e., male or female.
3. Patients listed for abdominal surgeries
4. American Society of Anesthesiologists (ASA) the status of I or II

Exclusion Criteria:

1. Patients with history of drug allergy.
2. Patients with liver disease, kidney disease, cardiac disease or sickle cell anemia,severe preeclampsia CNS disorder on history. Clinical and laboratory assessment
3. American Society of Anesthesiologists (ASA status III or IV)
4. Patients with morbid obesity 5, Raynaud's disease

6. Patients on adrenoceptor agonists or antagonists or narcotics before the operation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-10-25 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Post op Analgesia Effectiveness | Up to 24 hours
  Duration of Post Op Analgesia

SECONDARY OUTCOMES:
Opioid sparing Effect | 24 hours
  Total opioid consumption in mg/24hrs

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Riaz, MD, Study Director — Sahiwal medical college sahiwal
Locations (1):
- Sahiwal Medical College, Sāhīwāl, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Date will be available on request after completion of study i.e. February 2026
Supporting Information: Study Protocol, SAP, ICF
Time Frame: February 2026